CLINICAL TRIAL: NCT07325955
Title: Effect of Long Term Trimetazidine Treatment on Myocardial Final Fibrosis for Acute Myocardial Infarction
Brief Title: Effect of Long Term Trimetazidine Treatment on Final Myocardial Fibrosis for ST Eleviation Myocardial Infarction
Acronym: Easy
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, MD, Chinese PLA General Hospital
Other Study IDs: TMZAMI002; SF2020-2-5012 (Other: Chinese PLA General Hospital)
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: ST Elevation Myocardial Infarction (STEMI)
Keywords: Acute myocardial infarction; Trimetazidine; Metabolic therapy
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trimetazidine treatment group: Patients with trimetazidine treatment
- Control group: Patients without Trimetazidine treatment

SUMMARY:
Trimetazidine is a agent promoting glucose utilization by limiting fatty-acid oxidation.Trimetazidine could improve cardiac function in patients with ischemic heart disease. We aimed to explore effect of Trimetazidine on final myocardial fibrosis for patients with ST-elevation myocardial infarction (STEMI) in real world clinical practice. In this observational study, we investigated the effect of long-term treatment with trimetazidine on the final extent of myocardial fibrosis measured by cardiac magnetic resonance 6 months after infarction in real world clinical practice.

DETAILED DESCRIPTION:
This study is an prospective observational real-world clinical research. We evaluated the effect of long term trimetazidine treatment after the primary percutaneous coronary intervention (PCI), the myocardial infarction size in STEMI patients could be further reduced by metabolic regulation therapy. This study contributes to the development of standardized treatment procedure for STEMI patients.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed STEMI patients within one day after reperfusion threapy; Have performed the primary PCI procedure; Sign the informed consent form for this cohort study

Exclusion Criteria:

Mechanical complications; Cardiogenic shock; Malignant tumors, severe infection, hepatic or renal failure, respiratory failure, or other short-term progressive diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants were recruited from the Chinese PLA general hospital in Beijing
Sampling Method: Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
myocardial fibrosis measured by cardiac magnetic resonance imaging | 6 months after infarction
  Delayed enhancement of cardiac magnetic resonance imaging showed the myocardial fibrosis after infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA general hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Demirelli S, Karakelleoglu S, Gundogdu F, Tas MH, Kaya A, Duman H, Degirmenci H, Hamur H, Simsek Z. The Impact of Trimetazidine Treatment on Left Ventricular Functions and Plasma Brain Natriuretic Peptide Levels in Patients with Non-ST Segment Elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention. Korean Circ J. 2013 Jul;43(7):462-7. doi: 10.4070/kcj.2013.43.7.462. Epub 2013 Jul 31. PMID 23964292
- [Result] Shehata M. Cardioprotective Effects of Oral Trimetazidine in Diabetic Patients With Anterior Wall Myocardial Infarction Treated with Thrombolysis. Cardiol Res. 2014 Apr;5(2):58-67. doi: 10.14740/cr330w. Epub 2014 May 15. PMID 28392876
- [Result] Li R, Tang X, Jing Q, Wang Q, Yang M, Han X, Zhao J, Yu X. The effect of trimetazidine treatment in patients with type 2 diabetes undergoing percutaneous coronary intervention for AMI. Am J Emerg Med. 2017 Nov;35(11):1657-1661. doi: 10.1016/j.ajem.2017.05.024. Epub 2017 May 23. PMID 28587952
- [Result] Li Y, Wang D, Hu C, Zhang P, Zhang D, Qin S. Efficacy and Safety of Adjunctive Trimetazidine Therapy for Acute Myocardial Infarction: A Systematic Review and Meta-Analysis. Cardiology. 2016;135(3):188-195. doi: 10.1159/000446640. Epub 2016 Jul 15. PMID 27415810
- [Result] Banach M, Rysz J, Goch A, Mikhailidis DP, Rosano GM. The role of trimetazidine after acute myocardial infarction. Curr Vasc Pharmacol. 2008 Oct;6(4):282-91. doi: 10.2174/157016108785909788. PMID 18855716
- [Result] El-Kady T, El-Sabban K, Gabaly M, Sabry A, Abdel-Hady S. Effects of trimetazidine on myocardial perfusion and the contractile response of chronically dysfunctional myocardium in ischemic cardiomyopathy: a 24-month study. Am J Cardiovasc Drugs. 2005;5(4):271-8. doi: 10.2165/00129784-200505040-00006. PMID 15984909
- [Result] Kim JS, Kim CH, Chun KJ, Kim JH, Park YH, Kim J, Choi JH, Lee SH, Kim EJ, Yu DG, Ahn EY, Jeong MH. Effects of trimetazidine in patients with acute myocardial infarction: data from the Korean Acute Myocardial Infarction Registry. Clin Res Cardiol. 2013 Dec;102(12):915-22. doi: 10.1007/s00392-013-0611-0. Epub 2013 Aug 28. PMID 23982468
- [Result] Bonello L, Sbragia P, Amabile N, Com O, Pierre SV, Levy S, Paganelli F. Protective effect of an acute oral loading dose of trimetazidine on myocardial injury following percutaneous coronary intervention. Heart. 2007 Jun;93(6):703-7. doi: 10.1136/hrt.2006.107524. Epub 2007 May 8. PMID 17488771
- [Result] Fragasso G, Palloshi A, Puccetti P, Silipigni C, Rossodivita A, Pala M, Calori G, Alfieri O, Margonato A. A randomized clinical trial of trimetazidine, a partial free fatty acid oxidation inhibitor, in patients with heart failure. J Am Coll Cardiol. 2006 Sep 5;48(5):992-8. doi: 10.1016/j.jacc.2006.03.060. Epub 2006 Aug 17. PMID 16949492
- [Result] Singh D, Oladimeji-Salami J, Akindele AJ. New insights on pharmacological and therapeutic potentials of trimetazidine beyond anti-anginal drug: A comprehensive review. Eur J Pharmacol. 2024 Dec 15;985:177062. doi: 10.1016/j.ejphar.2024.177062. Epub 2024 Oct 19. PMID 39427862